CLINICAL TRIAL: NCT04445883
Title: Evaluating the Impact of a Volunteer Based Mealtime Assistance Program on the Nutritional Status of Patients at Joseph Brant Hospital in Ontario, Canada
Brief Title: Evaluating the Impact of the Eating Matters Program on the Nutritional Status of Medical Rehab Patients at Joseph Brant Hospital
Acronym: JBH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph Brant Hospital (Other)
Collaborators: Western University (Other)
Responsible Party: Principal Investigator, Diala Chayab, Clinical Dietitian, Joseph Brant Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JosephBrantH
Record Dates: First submitted 2020-05-15; First posted 2020-06-24 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Food Intake

STUDY DESIGN:
Intervention Model Description: The investigators will be evaluating patients' nutritional outcomes in units that have the Eating Matters Program available vs. similar units that do not have this program. Therefore, there will be two groups, Study Group A and Control Group B.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group A (Experimental): Study group A will include patients from the medical unit on 6S100 in addition to the Rehab units on 6N400/500. Participants in Study Group A will be receiving mealtime assistance from volunteers via the Eating Matters Program.
  Interventions: Behavioral: Feeding Assistance
- Control Group B (No Intervention): Control Group B will include participants from the Rehab Unit on 4N400 and the Medical unit on 6S200.

INTERVENTIONS:
Behavioral: Feeding Assistance — Patients will be receiving assistance during mealtimes. This includes assistance by opening packages, listing/explaining the food products on the tray, providing encouragement and companionship during mealtimes and directly feed patients.
  Arms: Study Group A

SUMMARY:
This research study will determine the impact of the Eating Matters Program on the nutritional status of elderly patients at Joseph Brant Hospital. The Eating Matters Program at Joseph Brant Hospital is a volunteer-based feeding assistance program that aims to improve patients' nutritional intake by providing assistance during mealtimes. As research on the impact of such programs on food intake is limited in Canada, this study will explore how the Eating Matters Program influences protein and energy intake of patients at Joseph Brant Hospital. Further, this study will explore if the hypothesized increase in protein and energy intake with the initiation of the Eating Matters Program is correlated with a decreased risk of malnutrition.

DETAILED DESCRIPTION:
We will be conducting a prospective open-label non-randomized controlled trial to evaluate patients' nutritional outcomes in units that have the Eating Matters Program available (Study Group A) vs. similar units that do not have this program (Control Group B), as this can provide useful data on the effectiveness of such programs in developing innovative prevention strategies to address hospital malnutrition.

A total sample size of eighty participants (40 in each group) will be included in this study from Medical and Rehabilitation units at Joseph Brant Hospital. Study group A will include patients from the medical unit on 6S100 in addition to the Rehab units on 6N400/500. Control Group B will include participants from the Rehab Unit on 4N400 and the Medical unit on 6S200. Baseline food intake data (including breakfast, lunch and dinner) will be gathered during a 2-day period for both Study Group A and Control Group B. Following the collection of baseline data, feeding assistance will then be provided to participants in the units that have the EMP program available (6S100 and 6N400/500). In addition, food intake will be recorded for a total of 6 days for both Study Group A, and Control Group B. Outcome measures including C-reactive protein and weight will be measured weekly. Following, a Subjective Global Assessment (SGA) will be completed and Hand Grip Strength will be recorded on days 1 and 18 as the literature shows that this is an appropriate timeframe to reassess these measures (Flood et al., 2014; Canadian Malnutrition Task Force, 2019). Energy and protein intake will then be calculated using visual estimation by completion of the My Meal Intake Tool, and the hospital's CBORD software. Further, to evaluate the success of the feeding assistance program, volunteers will distribute the feedback survey to patients, staff, family members or friends of participants. To prevent contamination from staff working on both sides, members of the research team will have a discussion with staff to explain that the study and potential benefits should not be discussed, as this may impact the research findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients 65 years and over admitted to Medicine and Rehabilitation units at Joseph Brant Hospital with an anticipated stay 10-14 days
* Patients with a Subjective Global Assessment score of B or C, and identified to require eating assistance
* Patients able to provide consent or have a Power of Attorney to do so on their behalf

Exclusion Criteria:

* Patients that are NPO status (nothing by mouth)
* Patients that require enteral or total parenteral feeding
* Palliative care patients
* Severe cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Dietary Intake | To assess a change from baseline to energy and protein intake post program initiation at the one and two week mark (+/-2days).
  Protein and Energy Intake

OTHER OUTCOMES:
Percent weight change | A change from baseline body weight at 1 week and 2 weeks marks (+/-2) days post the initiation of the Eating Matters Program (EMP).
  Participants' weight will be measured.
Handgrip strength | A change from baselines in handgrip measure at 1 and 2 weeks marks (+/-2 days) post the initiation of EMP.
  Handgrip strength measured using hand dynamometers.
C-Reactive Protein | A change from baselines CRP at 1 week and 2 weeks marks (+/-2 days) post the initiation of EMP.
  C-Reactive Protein will be measured via routine lab work.
Eating Matters Program Feedback | This will be measured on day 19 (+/-2 days) (total study period for each participant).
  Perceptions of program implementation and Barriers to food intake will be evaluated via feedback forms.
Length of stay | This data will be gathered on day 120 (+/-2days), upon completion of the study.
  Unit Specific Measure
Mortality rate | This data will be gathered on day 120 (+/- 2days), upon completion of the study.
  Unit Specific Measure
Re-admission rate | This data will be gathered on day 120 (+/- 2 days), upon completion of the study.
  Unit Specific Measure

CONTACTS AND LOCATIONS:
Overall Officials: Latifa Ahmadi, PhD, Study Chair — Western University
Locations (1):
- Joseph Brant Hospital, Burlington, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The sponsor will comply with data sharing processes according to local laws and regulations. Aggregate study results will be reported on clinicaltrials.gov. Anonymized study IPD can only be shared upon request from a regulator, an ethics committee board or by a healthcare professional for future research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD and any additional supporting information will become available starting 6months post-study publications for a period of 2-5 years.
Access Criteria: IPD can only be shared upon request from a regulator, an ethics committee board or by a healthcare professional for future research purposes. The study sponsor and principal investigator will be responsible to review requests in accordance with local regulations and institutional policies.

REFERENCES:
- [Background] Allard JP, Keller H, Teterina A, Jeejeebhoy KN, Laporte M, Duerksen DR, Gramlich L, Payette H, Bernier P, Davidson B, Lou W. Lower handgrip strength at discharge from acute care hospitals is associated with 30-day readmission: A prospective cohort study. Clin Nutr. 2016 Dec;35(6):1535-1542. doi: 10.1016/j.clnu.2016.04.008. Epub 2016 Apr 13. PMID 27155939
- [Background] Allard JP, Keller H, Jeejeebhoy KN, Laporte M, Duerksen DR, Gramlich L, Payette H, Bernier P, Davidson B, Teterina A, Lou W. Decline in nutritional status is associated with prolonged length of stay in hospitalized patients admitted for 7 days or more: A prospective cohort study. Clin Nutr. 2016 Feb;35(1):144-152. doi: 10.1016/j.clnu.2015.01.009. Epub 2015 Jan 21. PMID 25660316
- [Background] Barker LA, Gout BS, Crowe TC. Hospital malnutrition: prevalence, identification and impact on patients and the healthcare system. Int J Environ Res Public Health. 2011 Feb;8(2):514-27. doi: 10.3390/ijerph8020514. Epub 2011 Feb 16. PMID 21556200
- [Background] Bharadwaj S, Ginoya S, Tandon P, Gohel TD, Guirguis J, Vallabh H, Jevenn A, Hanouneh I. Malnutrition: laboratory markers vs nutritional assessment. Gastroenterol Rep (Oxf). 2016 Nov;4(4):272-280. doi: 10.1093/gastro/gow013. Epub 2016 May 11. PMID 27174435
- [Background] Curtis LJ, Valaitis R, Laur C, McNicholl T, Nasser R, Keller H. Low food intake in hospital: patient, institutional, and clinical factors. Appl Physiol Nutr Metab. 2018 Dec;43(12):1239-1246. doi: 10.1139/apnm-2018-0064. Epub 2018 May 8. PMID 29738268
- [Background] Curtis LJ, Bernier P, Jeejeebhoy K, Allard J, Duerksen D, Gramlich L, Laporte M, Keller HH. Costs of hospital malnutrition. Clin Nutr. 2017 Oct;36(5):1391-1396. doi: 10.1016/j.clnu.2016.09.009. Epub 2016 Sep 19. PMID 27765524
- [Background] Eckert KF, Cahill LE. Malnutrition in Canadian hospitals. CMAJ. 2018 Oct 9;190(40):E1207. doi: 10.1503/cmaj.180108. No abstract available. PMID 30301744
- [Background] Edwards D, Carrier J, Hopkinson J. Assistance at mealtimes in hospital settings and rehabilitation units for patients (>65years) from the perspective of patients, families and healthcare professionals: A mixed methods systematic review. Int J Nurs Stud. 2017 Apr;69:100-118. doi: 10.1016/j.ijnurstu.2017.01.013. Epub 2017 Jan 30. PMID 28199923
- [Background] Flood A, Chung A, Parker H, Kearns V, O'Sullivan TA. The use of hand grip strength as a predictor of nutrition status in hospital patients. Clin Nutr. 2014 Feb;33(1):106-14. doi: 10.1016/j.clnu.2013.03.003. Epub 2013 Mar 27. PMID 23615623
- [Background] Marsik C, Kazemi-Shirazi L, Schickbauer T, Winkler S, Joukhadar C, Wagner OF, Endler G. C-reactive protein and all-cause mortality in a large hospital-based cohort. Clin Chem. 2008 Feb;54(2):343-9. doi: 10.1373/clinchem.2007.091959. Epub 2007 Dec 21. PMID 18156283
- [Background] Manning F, Harris K, Duncan R, Walton K, Bracks J, Larby L, Vari L, Jukkola K, Bell J, Chan M, Batterham M. Additional feeding assistance improves the energy and protein intakes of hospitalised elderly patients. A health services evaluation. Appetite. 2012 Oct;59(2):471-7. doi: 10.1016/j.appet.2012.06.011. Epub 2012 Jun 23. PMID 22735333
- [Background] Sandhaus S, Zalon ML, Valenti D, Dzielak E, Smego RA Jr, Arzamasova U. A volunteer-based Hospital Elder Life Program to reduce delirium. Health Care Manag (Frederick). 2010 Apr-Jun;29(2):150-6. doi: 10.1097/HCM.0b013e3181daa2a0. PMID 20436332
- [Background] Walton K, Williams P, Bracks J, Zhang Q, Pond L, Smoothy R, Tapsell L, Batterham M, Vari L. A volunteer feeding assistance program can improve dietary intakes of elderly patients--a pilot study. Appetite. 2008 Sep;51(2):244-8. doi: 10.1016/j.appet.2008.02.012. Epub 2008 Feb 17. PMID 18387692
- See also: Time to Eat Toolkit. Retrieved from Alberta Health Services — https://www.albertahealthservices.ca/nutrition/Page16003.aspx
- See also: Integrated Nutrition Pathway for Acute Care (INPAC) Implementation Toolkit — https://nutritioncareincanada.ca/sites/default/uploads/files/INPAC-Toolkit-FINAL-Dec5-2017.pdf
- See also: Assessment: SGA — https://nutritioncareincanada.ca/resources-and-tools/hospital-care-inpac/assessment-sga
- See also: Food Monitoring Tools — http://nutritioncareincanada.ca/sites/default/uploads/files/MAT-MITT-Tools_2017.pdf
- See also: Sample size calculation tool — http://www.sample-size.net/sample-size-means/
- See also: Tackling Malnutrition Resource — https://nutritioncareincanada.ca/prevention-and-awareness/healthcare-professionals-decision-makers